CLINICAL TRIAL: NCT05486377
Title: Efficacy and Safety of Remimazolam vs. Inhalational Anesthetics for General Anesthesia for the Ablation of Arrhythmia: Randomized Controlled Trial
Brief Title: Remimazolam vs Desflurane for General Anesthesia for Ablation of Arrhythmia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, In-Ae Song, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2205-757-001
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Remimazolam; Desflurane; Cryoablation; Arrhythmia; General Anesthesia
Keywords: Remimazolam; Desflurane; Arrhythmia; Cryoablation,heart; Cardiovascular disease
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): General anesthesia with remimazolam-remifentanil TIVA.
  Interventions: Drug: Remimazolam besylate
- Desflurane (No Intervention): General anesthesia with maintaining with desflurane (induction:PPF, remifentanil CIV)

INTERVENTIONS:
Drug: Remimazolam besylate — Remimazolam besylate TIVA
  Arms: Remimazolam

SUMMARY:
In anesthesia for ablation for cardiac arrhythmias, abrupt hemodynamic changes or fatal arrhythmias can be seen frequently. Remimazolam is a novel ultra-short acting benzodiazepine that provides good hemodynamic stability compared to conventional anesthetic agents. This study aims to investigate whether remimazolam reduces vasoactive agent use during cryo/radiofrequancy ablation under general anesthesia, compared to desflurane(RCT).

ELIGIBILITY:
Inclusion Criteria:

* =or > 20 years
* Admission for General anesthesia for RFCA or cryoablation procedure

Exclusion Criteria:

* No severe adverse effect history or hypersensitivity of benzodiazepines or its additives
* Acute alcoholic intoxication state
* Coma or shock state due to other condition than heart problem.
* Acute narrow-angle glaucoma

Ages: 20 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Vasopressor CIV | During anesthesia
  Vasopressor CIV or not
Hypotension event | During and after anesthesia
  Hypotension event
Vasopressor (total amount) | During anesthesia
  Norepinephrine equivalent dose

SECONDARY OUTCOMES:
Induction time | Induction
  Induction dose administration~LOC
Recovery time | Recovery
  Reversal agent administration~extubation
Adverse event | During and after anesthesia (~24hr)
  Adverse event (desaturation, vomiting, hypotension, bleeding, allergic or anaphylaxis, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university Bundang hospital, Seongnam, Province (optional), South Korea

REFERENCES:
- [Derived] Yim S, Choi CI, Park I, Koo BW, Oh AY, Song IA. Remimazolam to prevent hemodynamic instability during catheter ablation under general anesthesia: a randomized controlled trial. Can J Anaesth. 2024 Aug;71(8):1067-1077. doi: 10.1007/s12630-024-02735-z. Epub 2024 Apr 12. PMID 38609684